CLINICAL TRIAL: NCT00907322
Title: A Phase 1, Investigator- And Subject-Blind (Sponsor-Open), Randomized, Crossover, Placebo-Controlled Trial To Assess The Safety, Tolerability, And Pharmacokinetics Of Single, Ascending, Oral Doses Of Dimebon [PF-01913539] In Healthy Adult Subjects
Brief Title: A Phase 1 Trial To Assess The Safety And Pharmacokinetics Of Single, Ascending, Oral Doses Of Dimebon In Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: B1451036
Record Dates: First submitted 2009-05-20; First posted 2009-05-22 (Estimated); Last update posted 2009-07-22 (Estimated); Status verified 2009-07

CONDITIONS: Healthy Volunteers
Keywords: oral, single ascending doses; CYP2D6 metabolizer status; healthy subjects; safety, tolerability, pharmacokinetics
MeSH Terms: interventions — latrepirdine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dimbeon 20 mg (Experimental)
  Interventions: Drug: Dimebon
- Dimebon 40 mg (Experimental)
  Interventions: Drug: Dimebon
- Dimebon 60 mg (Experimental)
  Interventions: Drug: Dimebon
- Placebo (Experimental)
  Interventions: Drug: Dimebon

INTERVENTIONS:
Drug: Dimebon — Oral tablet; 20 mg Dimebon, single dose
  Arms: Dimbeon 20 mg
Drug: Dimebon — Oral tablet; 40 mg Dimebon, single dose
  Arms: Dimebon 40 mg
Drug: Dimebon — Oral tablet; 60 mg Dimebon, single dose
  Arms: Dimebon 60 mg
Drug: Dimebon — Oral tablet; placebo, single dose
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of Dimebon following single ascending doses. A formal single ascending dose study of this nature has not been performed to date in the Dimebon development program.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive.
* Subjects who display the CYP2D6 extensive, intermediate, ultra-rapid, or poor metabolizer statuses.

Exclusion Criteria:

* A known history of hypersensitivity or previous intolerance to Dimebon or other antihistamines.
* Subjects with any previous history of seizures, convulsions, epilepsy, or significant head injury.
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Physical/neurological examination findings, clinical safety laboratory assessments, 12-lead ECGs, vital sign measurements, and adverse event monitoring. | July 2009
Pharmacokinetic parameters: Cmax, Tmax, AUClast, AUCinf, half-life, CL/F and Vz/F. | July 2009

SECONDARY OUTCOMES:
Pharmacodynamics: results of a Drug Effect Questionnaire | once each arm

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1451036&StudyName=A%20Phase%201%20Trial%20To%20Assess%20The%20Safety%20And%20Pharmacokinetics%20Of%20Single%2C%20Ascending%2C%20Oral%20Doses%20Of%20Dimebon%20In%20Healthy%20Adults